CLINICAL TRIAL: NCT06875661
Title: Treatment of Adolescent Idiopathic Scoliosis with the Conservative Schroth Method: a Randomized Controlled Trial
Brief Title: Treatment of Adolescent Idiopathic Scoliosis with the Schroth Method
Acronym: SchrothMED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Novi Sad (Other)
Responsible Party: Principal Investigator, Dragan Marinkovic, Lead Investigator, University of Novi Sad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 49-02-04/2023-1
Record Dates: First submitted 2025-03-07; First posted 2025-03-13 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Idiopathic Scoliosis
Keywords: Schroth method; Adolescent idiopathic scoliosis; Cobb angle; Spine health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Schroth (Experimental): Schroth experimental group
  Interventions: Other: Schroth
- Control (No Intervention): Group of participants without Schroth method intervention

INTERVENTIONS:
Other: Schroth — Patients in the experimental group exercised for 90 minutes a day, three days a week. Schroth exercises were performed in an asymmetrical position to improve the symmetry of the trunk. These exercises include stretching, flexion, spinal lengthening, derotation, strengthening, and rotational breathing exercises. The respondents combined these exercises with everyday life activities. In the control group, subjects were taught Schroth exercises under the supervision of an authorized physiotherapist, and they were asked to practice the exercises as regularly as possible at home.
  Arms: Schroth

SUMMARY:
This study investigates the effectiveness of the Schroth method, a conservative physiotherapeutic approach, in the treatment of adolescent idiopathic scoliosis (AIS). AIS is a three-dimensional spinal deformity of unknown etiology that develops during growth, affecting 2-3% of the general population. While most cases are mild, some require medical intervention, including bracing or surgery. Conservative treatments, such as specific exercise programs, aim to slow progression, improve postural alignment, and enhance respiratory function. Among these, the Schroth method is widely recognized for its structured approach, emphasizing active three-dimensional posture correction, rotational breathing, and sensorimotor training.

This study was designed as a randomized, single-blind, parallel-group trial conducted at Scolio Centar in Novi Sad between March and August 2023. Ethical approval was obtained from the Faculty of Sports and Physical Education, University of Novi Sad, and informed consent was secured from participants' parents. Inclusion criteria comprised a confirmed AIS diagnosis, an age range of 10-18 years, a Cobb angle greater than 10°, and no prior surgical or alternative treatment. Exclusion criteria included contraindications for exercise, psychological disorders, neuromuscular diseases, or previous spinal surgeries.

The study involved 34 participants who were randomly assigned to two groups: an experimental group (EG), which underwent supervised Schroth therapy three times a week for eight weeks, and a control group (CG), which performed the same exercises independently at home. Baseline and post-intervention assessments included radiographic measurement of Cobb angle, ATR via scoliometer, respiratory function tests (VC, FVC, FEV1, FEV1/FVC ratio) using spirometry, and CE via manual measurement. Stratified randomization was used to balance the groups based on Cobb angle severity.

The Schroth exercise protocol included posture correction exercises, spinal stabilization drills, and targeted breathing techniques, supervised by a certified physiotherapist for the EG. The CG received initial instruction but performed the exercises independently at home.

DETAILED DESCRIPTION:
Adolescent idiopathic scoliosis (AIS) is a complex three-dimensional deformity of the spine that develops between 10 years of age and skeletal maturity. It is characterized by lateral curvature, vertebral rotation, and sagittal plane changes. Despite extensive research, the exact etiology remains unknown, though genetic factors are believed to play a significant role. AIS affects 2-3% of the general population, with 10% of diagnosed individuals requiring some form of intervention, and 0.1% progressing to surgical treatment. The primary concerns in AIS management include curve progression, respiratory dysfunction, postural imbalance, and potential pain syndromes.

Conservative treatments aim to prevent scoliosis progression, reduce spinal deformity, and improve overall function. The most commonly used conservative approaches include the Schroth method, the Scientific Exercise Approach to Scoliosis (SEAS), the Lyon method, and core stabilization exercises. The Schroth method, developed by Katharina Schroth in the 1920s and refined over decades, is a structured physiotherapeutic approach that combines active three-dimensional posture correction, rotational breathing, and postural awareness training. It is widely used to improve spinal alignment, muscular symmetry, and pulmonary function in AIS patients.

Several studies have demonstrated the benefits of Schroth exercises, showing improvements in Cobb angle, trunk rotation, and respiratory function. However, there is ongoing debate regarding the efficacy of supervised therapy compared to self-administered home-based programs. This study aims to determine the effectiveness of supervised Schroth exercises in AIS patients and compare outcomes between supervised and unsupervised intervention groups.

Study Design This study was a randomized, single-blind, 1:1 parallel-group trial conducted at Scolio Centar in Novi Sad between March and August 2023. Ethical approval was obtained from the Ethics Committee of the Faculty of Sports and Physical Education, University of Novi Sad. Written informed consent was obtained from the parents of all participants before enrollment.

Participants

A total of 34 participants (24 males, 10 females) aged 11-16 years with AIS were recruited. Inclusion criteria included:

Diagnosis of AIS Age between 10 and 18 years Cobb angle >10° Risser sign between 0 and 5 No prior scoliosis treatment, including bracing or surgery

Exclusion criteria included:

Contraindications for exercise (e.g., cardiovascular or orthopedic limitations) Neuromuscular diseases Psychological conditions interfering with participation Prior spinal surgery Randomization and Blinding Participants were randomly assigned to either the experimental group (EG) or the control group (CG) using stratified randomization based on Cobb angle severity. Allocation was performed using sealed envelopes. The primary investigator conducting assessments was blinded to group allocation to reduce bias.

Intervention The intervention lasted eight weeks and consisted of three weekly sessions of 90 minutes each for the EG, performed under the supervision of Schroth-certified physiotherapists. The CG received an initial supervised training session on Schroth exercises and was instructed to perform the same exercises at home without further supervision.

The Schroth method includes:

Postural correction: Active realignment of the spine to reduce scoliosis curvature Rotational breathing: Directing inhaled air towards concave regions of the thorax to enhance spinal symmetry Muscle activation and stabilization: Strengthening targeted muscle groups to support spinal correction

The Schroth exercise protocol consisted of:

Warm-up exercises (general mobilization and activation)

Specific scoliosis correction exercises, including:

Side bending in a sitting position Derotation exercises in supine and prone positions Shoulder counter-traction exercises Core stabilization drills Breathing exercises targeting lung expansion and thoracic mobility Final stretching and relaxation exercises Outcome Measures

Baseline and post-treatment assessments were conducted for the following outcomes:

Cobb Angle (°): Measured via standing anterior-posterior radiographs Angle of Trunk Rotation (ATR) (°): Assessed using a Bunnell scoliometer in the forward bending position Vital Capacity (VC) (L): Measured using a Spirolab portable spirometer Forced Vital Capacity (FVC) (L): Evaluated through spirometry Forced Expiratory Volume in One Second (FEV1) (L): Determined via spirometry FEV1/FVC Ratio: Expressed as a percentage to assess airway function Chest Expansion (CE) (cm): Measured manually at the sternum-xiphoid junction using a tape measure

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of idiopathic scoliosis; Age range of 10-18 years (adolescent); Cobb angle greater than 10; No other types of exercise, medical treatment.

Exclusion Criteria:

The existence of some contraindications for exercise, psychological problems, neuro-logical-muscular diseases; Previous spine surgery.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 34 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-10 (Actual)

PRIMARY OUTCOMES:
The Cobb angle | 8 weeks
  The Coob angle expressed in degrees, was obtained using a standard anterior-posterior standing radiograph of the complete spine .
Angle of trunk rotation | 8 weeks
  The angle of trunk rotation (ATR) was measured with a Bunnell scoliometer, in a forward bending standing position. The scoliometer was placed on the patient's back cen-trally over the spine. ATR is expressed in degrees.
Vital Capacity (VC) | 8 weeks
  Vital Capacity (VC) as pulmonary function measured using a Spirolab Portable spirometer (MIR, Italy). The measurement was performed in an upright position. The procedure for each out-come was repeated three times and the average was taken as the reference value. Values are expressed in liters.
Forced Vital Capacity (FVC) | 8 weeks
  Forced Vital Capacity (FVC) as pulmonary function measured using a Spirolab Portable spirometer (MIR, Italy) and present maximum amount of air a person can forcibly exhale after taking a deep breath The measurement was performed in an upright position. The procedure for each out-come was repeated three times and the average was taken as the reference value. Values in liters.
Forced Expiratory Volume in One Second (FEV1) | 8 weeks
  Forced Expiratory Volume in One Second (FEV1) is the amount of air a person can forcibly exhale in the first second of a forced breath after taking a deep inhalation. Measuring using a Spirolab Portable spirometer (MIR, Italy). The measurement was performed in an upright position. The procedure for each out-come was repeated three times and the average was taken as the reference value. Values are expressed in liters.
Chest expansion | 8 weeks
  Chest expansion was measured manually using a tape marked in millimeters. Chest expansion was measured at the junction between the xiphoid process and the body of the sternum and expressed in centimeters.

SECONDARY OUTCOMES:
Date of birth | 8 weeks
  The participant's date of birth is collected in order to calculate his age in years.
Height | 8 weeks
  The height of the subject is determined in meters.
Weight | 8 weeks
  The weight of the participants is analyzed in kilograms.
Gender | 8 weeks
  The sex of the participants is recorded at the start of the study.
Body Mass Index (BMI) | 8 weeks
  The participant's BMI is calculated from his height and weight.

CONTACTS AND LOCATIONS:
Overall Officials: Dragan Marinkovic, Msc, Principal Investigator — University of Novi Sad, Faculty of Sport and Physical Education
Locations (1):
- University of Novi Sad, Faculty of Sport and Physical Education, Novi Sad, Serbia

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in scoliosis. Data will be coded, with no PHI included. Approval of the request and execution of all applicable agreements are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Data obtained through this study may be provided to qualified researchers with academic interest in scoliosis and spine disorders.